CLINICAL TRIAL: NCT06725147
Title: Digital Mental Health and Well-Being
Brief Title: Elomia - Digital Mental Health and Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Melissa Hunt, PhD, Associate Director of Clinical Training, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 857217
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Symptoms of Depression and Anxiety; Perceived Stress
Keywords: Psychological Wellbeing; Digital Mental Health; Artificial Intelligence; College Students; Elomia
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elomia - Digital Mental Health Chatbot (Experimental): Participants randomized to Elomia will be expected to use the intervention at least once per week (for around 30 minutes) but are encouraged to use as needed/wanted. Elomia is a generative AI program that can respond to text the user types in with unique responses that are designed to address therapeutic targets like stress, anxiety, procrastination, feeling overwhelmed and so on. Elomia was "trained" by real therapists with expertise in cognitive-behavioral therapy who responded to many different real people typing about their concerns. Thus, Elomia can suggest a number of different evidence based therapeutic strategies and can help the user process negative feelings, think through problems, plan solutions, and trouble shoot things that might get in the way of implementing those strategies.
  Interventions: Behavioral: AI enabled wellness chatbot
- Penn Wellness Modules (Active Comparator): Participants randomized to the control condition will be expected to use the intervention at least once per week (for around 30 minutes) but are encouraged to use as needed/wanted. The control condition consists of a curated collection of digital wellness resources that are already available freely to Penn students, including tips on getting good sleep, learning center material on time management and procrastination, and so on. The resources will be accessed via a single website, but there is no interactive component.
  Interventions: Behavioral: Penn Digital Wellness Resources

INTERVENTIONS:
Behavioral: AI enabled wellness chatbot — Elomia uses generative AI to respond to user input about psychological stress and distress. It was trained on the responses of real therapists with expertise in cognitive-behavioral therapy. It provides an array of wellness interventions including exercises for calming; • exercises for falling asleep; • grounding techniques; • exercises to reduce anxiety; • breathing exercises; • exercises to improve self-esteem.
  Arms: Elomia - Digital Mental Health Chatbot
Behavioral: Penn Digital Wellness Resources — This active control intervention consists of a variety of digital wellness and stress management resources that are freely available to all Penn students.
  Arms: Penn Wellness Modules

SUMMARY:
This study is testing the acceptability and efficacy of an AI enabled mental health chatbot (Elomia) as a resource of college student wellness.

DETAILED DESCRIPTION:
Elomia is a generative AI program that can respond to text users type in with unique responses that are designed to address therapeutic targets like stress, anxiety, procrastination, feeling overwhelmed and so on. Elomia was "trained" by real therapists with expertise in cognitive-behavioral therapy who responded to many different real people typing about their concerns. Thus, Elomia can suggest a number of different evidence based therapeutic strategies and can help the user process negative feelings, think through problems, plan solutions, and trouble shoot things that might get in the way of implementing those strategies. Elomia's arsenal includes:

* exercises for calming;
* exercises for falling asleep;
* grounding techniques;
* exercises to reduce anxiety;
* breathing exercises;
* exercises to improve self-esteem. The algorithm determines the user's need for one or another type of help while communicating with the chatbot and suggests an exercise to ease their emotional state. Elomia is not a substitute for professional care, and will detect when a person needs something more than a chatbot and will suggest connecting with other resources. More information about Elomia can be found via this website: https://elomia.com/

The ultimate goal of this study is to explore whether a mental health chatbot is acceptable and can improve symptoms of depression, anxiety, stress, and promote general psychological well-being in college students. The investigators will compare Elomia to a curated collection of digital wellness resources that are typically provided to students at our University.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student at the University of Pennsylvania.
* At least 18 years of age.

Exclusion Criteria:

* Severe depression or suicidality as indicated by Beck Depression Inventory score of >= 30, and/or a score of 2 or 3 on the Item (the suicide item) of the Beck Depression Inventory

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | Baseline and 4 week follow-up
  Self-report inventory of depressive symptoms Scores range from 0 to 63. Higher scores indicate more severe (worse) depressive symptoms.
GAD 7 | Baseline and 4 week follow-up
  Self-report inventory of symptoms of anxiety. Scores range from 0 to 21. Higher scores indicate more severe (worse) symptoms of anxiety.
Perceived Stress Scale | Baseline and 4 week follow-up
  Self-report questionnaire of perceived stress. Scores range from 0 to 40. Higher scores indicate more severe (worse) perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa G Hunt, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
To protect participant confidentiality

REFERENCES:
- See also: Elomia company website — https://elomia.com/